

### STATISTICAL ANALYSIS PLAN

**Study Title:** A Prospective, Open-Label, Multicenter, Phase 2 Trial to

Evaluate the Safety and Efficacy of the Combination of Tirabrutinib (GS-4059) and Idelalisib with and without Obinutuzumab in Subjects with Chronic Lymphocytic

Leukemia

Name of Test Drug: Tirabrutinib (GS-4059)

Study Number: GS-US-401-1958

**Protocol Version (Date):** Amendment 6 (28 May 2020)

**Analysis Type:** Final Analysis

**Analysis Plan Version:** Version 2.0

**Analysis Plan Date:** 16 February 2021

Analysis Plan Author: PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| STA | TISTIC | AL ANALYSIS PLAN | 1 |
|---|---|---|---|
| TAB | BLE OF | CONTENTS | 2 |
| LIST | Γ OF TA | BLES | 4 |
| | | BBREVIATIONS | |
| 1. | INTRO | DDUCTION | |
| | 1.1. | Study Objectives | |
| | 1.2. | Study Design | |
| | 1.3. | Sample Size and Power | |
| 2. | TYPE | OF PLANNED ANALYSIS | 10 |
| | 2.1. | Interim Analysis | 10 |
| | 2.2. | Final Analysis | |
| | 2.3. | Follow-up Analysis | 10 |
| 3. | GENEI | RAL CONSIDERATIONS FOR DATA ANALYSES | 11 |
| | 3.1. | Analysis Sets | 11 |
| | 5.1. | 3.1.1. All Enrolled Analysis Set | |
| | | 3.1.2. Full Analysis Set. | |
| | | 3.1.3. Safety Analysis Set | |
| | | CCI | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates | |
| | 3.4. | Examination of Subject Subgroups | |
| | 3.5.<br>3.6. | Multiple Comparisons | |
| | 3.0. | 3.6.1. Missing Data | |
| | | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | 13 |
| | 3.8. | Analysis Visit Windows | |
| | | 3.8.1. Definition of Study Day | |
| | | 3.8.2. Analysis Visit Windows | 14 |
| | | 3.8.2.1. Analysis Visit Windows for Primary/Secondary Efficacy | 1.5 |
| | | Endpoints | 15 |
| | | Window | 15 |
| 4. | SUBJE | CT DISPOSITION | 16 |
| | 4.1. | Subject Enrollment and Disposition | |
| | 4.1. | Extent of Study Drug Exposure and Adherence. | |
| | 7.2. | 4.2.1. Duration of Exposure to Study Drug | |
| | | 4.2.2. Adherence to Study Drug | |
| | 4.3. | Protocol Deviations | |
| | 4.4. | Assessment of COVID-19 Impact | |
| | | 4.4.1. Study Drug or Study Discontinuation Due to COVID-19 | |
| | | 4.4.2. Protocol Deviations Due to COVID-19 | |
| | | 4.4.3. Missed and Virtual Visits Due to COVID-19 | 19 |
| 5. | BASEI | INE CHARACTERISTICS | 20 |
| | 5.1. | Demographics | 20 |
| | 5.2. | Other Baseline Characteristics | |

| 5.3.<br>5.4. | | Historyti-cancer Therapy | |
|---|---|---|---|
| | | ALYSES | |
| 6.1. | | Efficacy Endpoint | |
| 0.1. | 6.1.1. | Definition of the Primary Efficacy Endpoint | |
| | 6.1.2. | Analysis of the Primary Efficacy Endpoint | |
| 6.2. | | ry Efficacy Endpoints | |
| 0.2. | 6.2.1. | Rates of CR/BM MRD- and CR/PB MRD- at Week 25 | |
| | 6.2.2. | ORR at Week 25 | |
| CCI | ſ | | |
| 6.4. | The second second | From Protocol-Specified Efficacy Analyses | |
| | 6.4.1. | ORR Time to Clinical Response CCI per Clinical Response Assessment | 27 |
| | 6.4.2. | Time to Clinical Response GCT per Clinical Response Assessment | 27 |
| SAFE | TY ANAL | LYSES | 29 |
| 7.1. | Adverse | Events and Deaths | 29 |
| | 7.1.1. | Adverse Event Dictionary | |
| | 7.1.2. | Adverse Event Severity | |
| | 7.1.3. | Relationship of Adverse Events to Study Drug | |
| | 7.1.4. | Serious Adverse Events | |
| | 7.1.5. | Treatment-Emergent Adverse Events | 29 |
| | | 7.1.5.1. Definition of Treatment-Emergent Adverse Events | |
| | | 7.1.5.2. Incomplete Dates | 30 |
| | 7.1.6. | Summaries of Adverse Events and Deaths | 30 |
| | | 7.1.6.1. Summaries of AE Incidence by Severity | 30 |
| | 7.1.7. | Adverse Events of Interest. | 32 |
| 7.2. | Laborato | ory Evaluations | 33 |
| | 7.2.1. | Summaries of Numeric Laboratory Results | |
| | 7.2.2. | Graded Laboratory Values | |
| | | 7.2.2.1. Treatment-Emergent Laboratory Abnormalities | |
| | | 7.2.2.2. Summaries of Laboratory Abnormalities | |
| | 7.2.3. | Liver-related Laboratory Evaluations | |
| | 7.2.4. | Shifts Relative to the Baseline Value | |
| 7.3. | 200/1 | eight and Vital Signs | |
| 7.4. | | d Concomitant Medications | |
| | 7.4.1.<br>7.4.2. | Prior Medications | |
| 75 | | ardiogram Results | |
| 7.5. | 7.5.1. | Investigator Electrocardiogram Assessment | |
| | 7.5.2. | Corrected QT Intervals | |
| | 7.5.3. | PR and QRS Intervals | |
| 7.6. | | afety Measures | |
| 7.7. | | From Protocol-Specified Safety Analyses | |

| 9. | REFERENCES. | | 40 |
|-----|--------------|------------------------------------------------|----|
| 11. | SAP REVISION | | 42 |
| 12. | APPENDICES | | 43 |
| | | LIST OF TABLES | |
| | Table 1-1. | 90% Confidence Intervals at Different CR Rates | 9 |

#### LIST OF ABBREVIATIONS

AE adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase

ATC Anatomical Therapeutic Chemical BLQ below the limit of quantitation

BM bone marrow BMI body mass index

CCR clinical complete response

CI confidence interval

CLL chronic lymphocytic leukemia

CPR clinical partial response
CR complete remission

CR/BM complete remission with bone marrow minimal residual disease negativity (<10<sup>-4</sup> CLL cells

MRD- present)

CR/PB complete remission with peripheral minimal residual disease negativity (<10-4 CLL cells

MRD- present)

CRi complete remission with incomplete recovery of the bone marrow

CRF case report form
CSR clinical study report

CTCAE Common Toxicity Criteria for Adverse Events

CCI

ECG electrocardiogram
EOT End of Treatment
FAS Full Analysis Set
HLT high-level term
ID identification

IWCLL International Workshop on CLL
IWRS Interactive Web Response System

LLT lower-level term
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

NLP Natural Language Processing

nPR nodular partial response
ORR overall response rate

CCI Overall respo

PB peripheral blood PD progressive disease

CCI

PP per protocol

PR partial response

PR-L partial response with lymphocytosis

PT preferred term

Q1, Q3 first quartile, third quartile

QRS electrocardiographic deflection between the beginning of the Q wave and termination of the

S wave representing time for ventricular depolarization

QT electrocardiographic interval between the beginning of the Q wave and termination of the

T wave representing the time for both ventricular depolarization and repolarization to occur

QTc QT interval corrected for heart rate

QTcF QT interval corrected for heart rate using Fridericia's formula

RR electrocardiographic interval representing the time measurement between the R wave of one

heartbeat and the R wave of the preceding heartbeat

SAP statistical analysis plan

SD stable disease StD standard deviation

SI (units) international system of units

SOC system organ class

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings

CCI

ULN upper limit of normal VR ventricular rate

WHO World Health Organization

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the synoptic clinical study report (CSR) for Study GS-US-401-1958. This SAP is based on the study protocol amendment 6 dated 28 May 2020 and the electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

### 1.1. Study Objectives

The primary objective of this study is:

 To determine the preliminary efficacy of the combination of tirabrutinib and idelalisib with obinutuzumab in subjects with relapsed or refractory chronic lymphocytic leukemia (CLL)

The secondary objective of this study is:

 To evaluate the safety and tolerability of the combination of tirabrutinib and idelalisib with and without obinutuzumab



### 1.2. Study Design

This is a Phase 2, prospective, open-label, multicenter trial to evaluate the safety and efficacy of the combination of tirabrutinib and idelalisib with and without obinutuzumab in subjects with relapsed or refractory CLL.

Eligible subjects will be randomized in a 1:1 manner to one of the following two arms, stratified by the presence of 17p deletion/TP53 mutation (del17p/TP53mut) in CLL cells:

- Arm A: tirabrutinib + idelalisib
- Arm B: tirabrutinib + idelalisib + obinutuzumab

With Amendment 3, randomization was discontinued. All subsequent subjects will be enrolled into Arm B.

# **Duration of Treatment:**

Tirabrutinib 80 mg and idelalisib 100 mg will be self-administered orally once daily. Dosing of both agents will begin on Week 1 Day 1 of the study and thereafter continue for up to 104 weeks in the absence of disease progression, unacceptable toxicity, or documentation of complete remission (CR) with bone marrow minimal residual disease (MRD) negativity (CR/BM MRD-). If CR/BM MRD- is documented on study, treatment will stop after the earlier of:

- i) an additional 3 months of therapy or
- ii) 104 weeks of total treatment.

Obinutuzumab will be administered as 8 intravenous infusions of 1000 mg each over 21 weeks. A test dose of 100 mg will be administered on Week 1 Day 1. If this dose is tolerated, the remainder of the full dose may be subsequently administered on Day 1. Alternatively, the remaining 900 mg will be administered on Day 2. Subsequent infusions will be administered on Week 2 Day 1, Week 3 Day 1, Week 5 Day 1 and then every 4 weeks through Week 21.

This study will continue to monitor subjects for up to 30 days post end of treatment, or up to Week 25 should a subject discontinue treatment prior to Week 25 for reasons other than disease progression.

#### **Efficacy Assessment Schedule:**

Tumor response assessment per modified International Workshop on CLL (IWCLL) 2008 criteria will be performed at the Week 25 visit, with evaluation of areas affected by CLL during the screening evaluation. During the treatment phase, additional response assessment per IWCLL 2008 criteria may be performed as clinically indicated.

Clinical response based on physical exam, laboratory parameters and presence of B-symptoms will be performed every 4 weeks until Week 33 Day 1 (except for Week 25) and then every 12 weeks starting Week 33 until Week 105 following the modified IWCLL 2008 criteria, with the exception of lymphadenopathy, hepatomegaly, splenomegaly, and bone marrow.

Bone marrow MRD will be assessed at Week 25. Additional bone marrow MRD may be assessed as clinically indicated. Peripheral blood MRD will be assessed on Day 1 of Weeks 1, 13, 25, 33, 45, 105, and End of Treatment (EOT). EOT collection is not needed for subjects who complete the Week 105 visit.

The Schedule of Assessments is located in Appendix 1.

# 1.3. Sample Size and Power

The primary goal of this study is to evaluate the efficacy of the combination of tirabrutinib and idelalisib with obinutuzumab in relapsed and refractory CLL. The evaluation will be based on the estimation of the CR rate (including CR and CR with incomplete recovery of the bone marrow (CRi)) and its corresponding exact confidence interval. Approximately 30 subjects will be enrolled into Arm B, which will result in the 90% confidence interval (CI) of the observed CR rate to be within ±17.0%. The 90% CI for a given observed CR rate is provided in Table 1-1.

Table 1-1. 90% Confidence Intervals at Different CR Rates

| Sample Size | Observed CR Rate | 90% Confidence Interval<br>using Clopper-Pearson Method |
|---|---|---|
| 30 | 20% | (9.1%, 35.7%) |
| 30 | 30% | (16.6%, 46.5%) |
| 30 | 40% | (25.0%, 56.6%) |
| 30 | 50% | (33.9%, 66.1%) |
| 30 | 60% | (43.4%, 75.1%) |

With Amendment 3, randomization was discontinued. All subsequent subjects will be enrolled to Arm B. A total of approximately 6 subjects in Arm A and 30 subjects in Arm B will be enrolled, thus the total sample size for the study will be approximately 36 subjects.

# 2. TYPE OF PLANNED ANALYSIS

# 2.1. Interim Analysis

No formal interim analysis is planned.

This study does not have a data monitoring committee (DMC). Therefore, no analyses will be conducted for the DMC.

# 2.2. Final Analysis

After all subjects have discontinued/completed the study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized, the final analysis of the data will be performed.

# 2.3. Follow-up Analysis

No follow-up analysis is planned.

### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (StD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-subject listings will be presented for all subjects in the All Enrolled Analysis Set and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within the subject. The treatment group to which subjects were randomized/initially assigned will be used in the listings. Age, sex at birth, race, and ethnicity for each subject will be presented in the listings, as space permits.

# 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of subjects eligible for inclusion will be summarized by treatment group.

A listing of reasons for exclusion from analysis sets will be provided by subject.

This study was initially designed as a randomized study. With Amendment 3, randomization was discontinued, and all subsequent subjects will be enrolled into Arm B. There is no intention to compare the treatments, so intent-to-treat Analysis Set will not be used; instead, All Enrolled Analysis Set defined in Section 3.1.1 and Full Analysis Set defined in Section 3.1.2 will be used.

# 3.1.1. All Enrolled Analysis Set

All Enrolled Analysis Set includes all subjects who received a study subject identification number in the study after screening.

# 3.1.2. Full Analysis Set

The Full Analysis Set (FAS) includes all subjects who received at least 1 dose of any study drug with treatment group designated according to the planned treatment. This is the primary analysis set for efficacy analyses.

# 3.1.3. Safety Analysis Set

The Safety Analysis Set includes all subjects who took at least 1 dose of study drug. This is the primary analysis set for safety analyses.



# 3.2. Subject Grouping

For analyses based on FAS, subjects will be grouped according to the treatment they are assigned to at randomization or enrollment. For analyses based on the Safety Analysis Set, subjects will be grouped according to the actual treatment received. The actual treatment received will differ from the treatment assigned at randomization or enrollment only when their actual treatment differs from assigned treatment for the entire treatment duration.



#### 3.3. Strata and Covariates

Subjects will be randomly assigned to treatment groups via the interactive web response system (IWRS) in a 1:1 ratio using a stratified randomization schedule. Stratification will be based on the presence of del17p/TP53mut in CLL cells. If there are discrepancies in stratification factor values between the IWRS and the clinical database, the values recorded in the clinical database will be used for analyses.

With Amendment 3, randomization was discontinued. All subsequent subjects were enrolled into Arm B. There is no intention to compare the treatments. No covariates will be included in efficacy analyses.

### 3.4. Examination of Subject Subgroups

Primary and secondary efficacy endpoints will be examined in the subgroups based on randomization stratification factor (either del17p or TP53mut versus neither del17p nor TP53mut) for each arm. CCI

#### 3.5. Multiple Comparisons

Not applicable.

#### 3.6. Missing Data and Outliers

### 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 4.2.1. The handling of missing or incomplete dates for CLL diagnosis is described in Section 5.3; for prior anti-cancer therapy in Section 5.4, for new anti-cancer therapy in Section 6.3.2, for death in Section 6.3.1, for AE onset in Section 7.1.5.2, and for prior and concomitant medications in Section 7.4.

#### **3.6.2. Outliers**

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be conducted. All data will be included in the data analysis.

# 3.7. Data Handling Conventions and Transformations

The following conventions will be used for the imputation of date of birth when it is partially missing or not collected:

- If only month and year of birth is collected, then "15" will be imputed as the day of birth
- If only year of birth is collected, then "01 July" will be imputed as the day and month of birth
- If year of birth is missing, then date of birth will not be imputed. In general, age collected at Day 1 (the first dosing date of study drug) (in years) will be used for analyses and presented in listings. If age at Day 1 is not available for a subject, then age derived based on date of birth and the Day 1 visit date will be used instead. If an enrolled subject was not dosed with any study drug, the randomization or enrollment date will be used instead of the Day 1 visit date. For screen failures, the date the first informed consent was signed will be used for the age derivation. Age required for longitudinal and temporal calculations and analyses (eg, estimates of creatinine clearance, age at date of AE) will be based on age derived from date of birth and the date of the measurement or event, unless otherwise specified.

Non-PK data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "< x" (where x is considered the LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used to calculate summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used to calculate summary statistics.
- A value that is 1 unit above the LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "> x" (where x is considered the LOQ). Values with decimal points will follow the same logic as above.
- The LOQ will be used to calculate descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the LOQ).

If methods based on the assumption that the data are normally distributed are not adequate, analyses may be performed on transformed data or nonparametric analysis methods may be used, as appropriate.



# 3.8. Analysis Visit Windows

### 3.8.1. Definition of Study Day

Study day will be calculated from the first dosing date of study drug and derived as follows:

- For postdose study days: Assessment Date First Dosing Date + 1
- For days prior to the first dose: Assessment Date First Dosing

Therefore, study day 1 is the day of first dose of study drug administration.

### 3.8.2. Analysis Visit Windows

The nominal visit as recorded on the CRF will be used when data are summarized by visit. Any data relating to unscheduled visits will not be assigned to a particular visit or time point. However, the following exceptions will be made:

- An unscheduled visit prior to the first dosing of study drug may be included in the calculation of the baseline value, if applicable.
- Unscheduled visits after the first dosing of study drug will be included in determining the maximum postbaseline toxicity grade.

# 3.8.2.1. Analysis Visit Windows for Primary/Secondary Efficacy Endpoints

The analysis windows for Week 25 response assessment and Week 25 MRD assessment are defined as 24×7±28 days (inclusive) starting from first dose.

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple valid, nonmissing measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline, the last nonmissing value on or prior to the first dosing date of study drug will be selected, unless specified differently. If there are multiple records with the same time or no time recorded on the same day, the baseline value will be the average of the measurements for continuous data, or the measurement with the lowest severity (eg, normal will be selected over abnormal for safety electrocardiogram [ECG] findings) for categorical data.
- For postbaseline values:
  - The record closest to the nominal day for that visit will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the average will be taken for continuous data and the worse severity will be taken for categorical data, unless otherwise specified.

# 4. SUBJECT DISPOSITION

### 4.1. Subject Enrollment and Disposition

A summary of subject enrollment will be provided by treatment group for each investigator and overall. The summary will present the number and percentage of subjects enrolled. For each column, the denominator for the percentage calculation will be the total number of subjects analyzed for that column.

A listing of subjects with discrepancies in the value used for stratification assignment between the IWRS and the clinical database at the time of data finalization will be provided.

A summary of subject disposition will be provided by treatment group. This summary will present the number of subjects screened, the number of subjects randomized or enrolled, the number of subjects who were randomized or enrolled but not dosed, and the number of subjects in each of the categories listed below by treatment group:

- Safety Analysis Set
- Tirabrutinib completion status
  - Completed study drug dosing as specified per protocol
  - Discontinued study drug dosing with reasons
- Idelalisib completion status
  - Completed study drug dosing as specified per protocol
  - Discontinued study drug dosing with reasons
- Obinutuzumab completion status
  - Completed study drug dosing as specified per protocol
  - Discontinued study drug dosing with reasons
- Study completion status
  - Completed the protocol-planned duration of the study
  - Discontinued the study with reasons

For the status of study drug and study completion and reasons for discontinuation, the number and percentage of subjects in each category will be provided. The denominator for the percentage calculation will be the total number of subjects in the All Enrolled Analysis Set corresponding to that column. In addition, a flowchart will be provided to depict the disposition.

The following by-subject listings will be provided by subject identification (ID) number in ascending order to support the above summary tables:

- Reasons for study drug or study discontinuation
- Reasons for screen failure (will be provided by screening ID number in ascending order)

### 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to study drug will be examined by assessing the total duration of exposure to study drug and the level of adherence to the study drug specified in the protocol.

### 4.2.1. **Duration of Exposure to Study Drug**

Total duration of exposure to study drug will be defined as last dosing date minus first dosing date plus 1, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). If the last study drug dosing date is missing, the latest date among the study drug end date, clinical visit date, laboratory sample collection date, and vital signs assessment date will be used.

The total duration of exposure to study drug will be summarized using descriptive statistics. For tirabrutinib and idelalisib, the number (ie, cumulative counts) and percentage of subjects exposed will be summarized by the following time periods:  $\geq 1$  day,  $\geq 1$  week,  $\geq 2$  weeks,  $\geq 3$  weeks,  $\geq 4$  weeks,  $\geq 6$  weeks,  $\geq 8$  weeks, every 4 weeks starting from 8 weeks to 32 weeks, and then every 12 weeks starting from 32 weeks until 104 weeks (if appropriate). For obinutuzumab, the number of infusions will be summarized using descriptive statistics. Summaries will be provided by treatment group for the Safety Analysis Set.

The number and percentage of subjects who have dose reduction or interruptions, and the reasons, will be summarized by treatment.

No formal statistical testing is planned.

#### 4.2.2. Adherence to Study Drug

The total amount of study drug administered (mg) will be summarized using descriptive statistics.

For tirabrutinib and idelalisib, the presumed total number of doses administered to a subject will be determined by the data collected on the drug accountability CRF using the following formula:

Total Amount of Study Drug Administered (mg) =

$$\left(\sum No. \text{ of Doses Dispensed} \times strength\right) - \left(\sum No. \text{ of Doses Returned} \times strength\right)$$

The level of on-treatment adherence to the study drug regimen will be determined by the total amount of study drug administered relative to the total amount of study drug expected to be administered during a subject's actual on-treatment period based on the study drug regimen. Investigator-prescribed interruption, reductions and escalations as specified in the protocol will be taken into account. If there are treatment periods that bottles are not returned or the return information is missing, these periods will be excluded from the on-treatment adherence calculation for both total amount of study drug administered and study drug expected to be administered. If subjects never returned any bottle, the adherence will be set as missing.

The level of on-treatment adherence will be expressed as a percentage using the following formula:

On-Treatment Adherence (%) = 
$$\left(\frac{\text{Total Amount of Study Drug Administered}}{\text{Study Drug Expected to be Administered on Treatment}}\right) \times 100$$

Descriptive statistics for the level of on-treatment adherence with the number and percentage of subjects belonging to adherence categories (eg, < 75% and  $\ge 75\%$ ) will be provided by treatment group for the Safety Analysis Set.

A by-subject listing of study drug administration and drug accountability will be provided separately by subject ID number (in ascending order) and visit (in chronological order).

#### 4.3. Protocol Deviations

Subjects who did not meet the eligibility criteria for study entry but enrolled in the study will be summarized regardless of whether they were exempted by the sponsor or not. The summary will present the number and percentage of subjects who did not meet at least 1 eligibility criterion and the number of subjects who did not meet specific criteria by treatment group based on the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects who did not meet at least 1 eligibility (inclusion or exclusion) criterion. The listing will present the eligibility criterion (or criteria if more than 1 deviation) that subjects did not meet and related comments, if collected.

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with important protocol deviations by deviation reason (eg, nonadherence to study drug, violation of select inclusion/exclusion criteria)

will be summarized by treatment group for the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects with important protocol deviation.

# 4.4. Assessment of COVID-19 Impact

This study was ongoing during the novel coronavirus (2019 nCOV [COVID-19]) pandemic, and the COVID-19 pandemic has caused a disruption in the regular visit schedules for this study. Some subjects were unable to attend onsite visits due to shelter in place guidelines, site closures, or other reasons. This section provides how to handle special situations due to COVID-19 in the analysis.

Adverse events (AEs) due to COVID-19 will be included in AE analyses if applicable. A bysubject listing of Adverse Events due to COVID-19 may be provided. The COVID-19 Standardized MedDRA Queries (SMQ) with Broad Scope in Appendix 2 will be implemented.

# 4.4.1. Study Drug or Study Discontinuation Due to COVID-19

A by-subject listing of reasons for premature study drug or study discontinuation due to COVID-19 will be created.

#### 4.4.2. Protocol Deviations Due to COVID-19

A by-subject listing will be provided for subjects with important protocol deviation related to COVID-19. A separate listing will be provided for subjects with non-important protocol deviation related to COVID-19.

#### 4.4.3. Missed and Virtual Visits Due to COVID-19

A by-subject listing of subjects with missed or virtual visits due to COVID-19 will be provided by subject ID number in ascending order .

Information regarding virtual or missed visits due to COVID-19 was collected as free text in the CRF comment fields. The determination of missing or virtual visits due to COVID-19 was done using Natural Language Processing (NLP) to search the CRF comment fields. A detailed explanation of the algorithm is given in Appendix 3.

### 5. BASELINE CHARACTERISTICS

# 5.1. Demographics

Subject demographic variables (ie, age, sex, race, and ethnicity) will be summarized by treatment group and overall using descriptive statistics for age, and using number and percentage of subjects for sex, race, and ethnicity. The summary of demographic data will be provided for FAS.

A by-subject demographic listing, including the informed consent date, will be provided by subject ID number in ascending order.

#### **5.2.** Other Baseline Characteristics

Other baseline characteristics include body weight (in kg), height (in cm), body mass index (BMI; in kg/m²), Eastern Cooperative Oncology Group (ECOG) Performance Status, CIRS (Cumulative Illness Rating Scale), fluorescence in situ hybridization (FISH) results, TP53 mutation status, and IGHV mutation status. These baseline characteristics will be summarized by treatment group and overall using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables. The summary of baseline characteristics will be provided for FAS. No formal statistical testing is planned.

A by-subject listing of other baseline characteristics will be provided by subject ID number in ascending order.

# **5.3.** Medical History

Medical history will be collected at screening for disease-specific and general conditions (ie, conditions not specific to the disease being studied).

Disease-specific medical history will be summarized by treatment group and overall by the number and percentage of subjects with each prepopulated condition. The summary will be provided for FAS. Time since CLL diagnosis (years) will be calculated by (date of first dose of study drug – date of CLL diagnosis) / 365.25. Time since CLL diagnosis will be summarized using summary statistics for a continuous variable. Disease stage at diagnosis and at screening and cytogenetic risk group will be summarized using summary statistics for a categorical variable. No formal statistical testing is planned. A by-subject listing of disease-specific medical history will be provided by subject ID number in ascending order.

In deriving the time since CLL diagnosis, all partial dates of diagnosis and last regimen will be identified, and the partial dates will be imputed as follows:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month.
- Partial date will not be imputed if the year is missing.

General medical history data will not be coded, but will be listed only. A by-subject listing of general medical history will be provided by subject ID number in ascending order.

# 5.4. Prior Anti-cancer Therapy

Number of prior regimens, time since the completion of last regimen, and time since progression in the last regimen will be summarized by treatment group using descriptive statistics based on FAS. A partial completion date will be imputed using the algorithm defined in Section 5.3.

The regimens and prior therapies that the subjects received will be summarized. The last regimen subjects received prior to study entry and the best response and PD to the last regimen will be summarized.

Number of subjects who received prior radiation therapy and surgery will be listed.

### 6. EFFICACY ANALYSES

Efficacy analysis will be performed on FAS. The result summary will be provided by treatment group if not otherwise specified.

### 6.1. Primary Efficacy Endpoint

# 6.1.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint of this study is the rate of CR per modified IWCLL 2008 criteria {Hallek 2008} at Week 25, which is defined as the proportion of subjects who achieved CR/CRi at Week 25. Subjects who received anti-cancer therapy other than the study drug prior to achieving CR/CRi at Week 25, will be considered as nonresponders for CR/CRi and will be included in the denominator when calculating the CR rate at Week 25.

The analysis window of Week 25 response assessment is defined as  $24 \times 7 \pm 28$  days (inclusive) starting from first dose. This analysis window is extended from the visit window to capture the assessments outside the scheduled window. If there are multiple assessments within the analysis window, records will be chosen based on rules specified in Section 3.8.3.

# 6.1.2. Analysis of the Primary Efficacy Endpoint

The CR rate at Week 25 and the corresponding 2-sided 90% exact CIs based on Clopper-Pearson method will be presented.

# 6.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints are:

- Rate of CR with MRD negativity (<10-4) in bone marrow (CR/BM MRD-) at Week 25, defined as the proportion of subjects who achieved CR/CRi and also achieved BM MRD negativity at Week 25
- Rate of CR with MRD negativity (<10<sup>-4</sup>) in peripheral blood (CR/PB MRD-) at Week 25, defined as the proportion of subjects who achieved CR/CRi and also achieved PB MRD negativity at Week 25
- Overall response rate (ORR) at Week 25, defined as the proportion of subjects who achieved CR, CRi, partial response (PR), or PR with lymphocytosis at Week 25

The response assessment definition of each response category is based on Modified IWCLL 2008 criteria and PR includes nodular partial response (nPR).

The MRD response is assessed with four-color-flow cytometry (FACS) and MRD negativity is defined as one CLL cell per 10,000 leukocytes [0.01 %], ie, <10<sup>-4</sup>.

The analysis window of Week 25 response assessment is defined as 24×7±28 days(inclusive) starting from first dose. If there are multiple assessments within the analysis window, records will be chosen based on rules specified in Section 3.8.3.

#### 6.2.1. Rates of CR/BM MRD- and CR/PB MRD- at Week 25

Subjects who received anti-cancer therapy other than the study drug prior to achieving CR with MRD negativity at Week 25 will be considered as nonresponders and will be included in the denominators of the response rates.

The rates of CR/BM MRD- and CR/PB MRD- and the corresponding 2-sided 90% exact CIs based on Clopper-Pearson method will be presented.

#### 6.2.2. ORR at Week 25

When calculating ORR at Week 25, subjects who received anti-cancer therapy other than the study drug prior to achieving responses at Week 25, will be considered as nonresponders and will be included in the denominator.

ORR at Week 25 and the corresponding 2-sided 90% exact CIs based on Clopper-Pearson method will be presented.

A by-subject listing of overall response based on modified IWCLL 2008 criteria will be provided.

A by-subject listing of BM and PB MRD results will be provided.









# 6.4. Change From Protocol-Specified Efficacy Analyses

As understanding of clinical response and response per modified IWCLL 2008 criteria beyond week 25 are desired, the following endpoints not defined by protocol will also be analyzed:

- ORR, defined as the proportion of subjects achieving best overall response of CR, CRi, PR, or PR with lymphocytosis per Modified IWCLL 2008 criteria while on study
- Time to clinical response, defined as the interval from first dose of study drug to the date of the first clinical response which includes clinical complete response (CCR) and clinical partial response (CPR)



Clinical response assessment is a qualitative treatment response assessment based on physical exam, laboratory parameters and presence of B-symptoms performed every 4 weeks until Week 33 Day 1 and then at all scheduled visits thereafter following the modified IWCLL 2008 criteria, with the exception of lymphadenopathy, hepatomegaly, splenomegaly, and bone marrow. Clinical response categories are CCR, CPR, stable disease, and suspected progressive disease.

The date of disease progression will be the time point at which progression is first identified by relevant radiographic imaging data or clinical data.

#### 6.4.1. ORR

The analysis will be performed with data collected throughout the study. Subjects, who never achieved these responses or received anti-cancer therapy other than the study drug prior to achieving responses, will be considered as nonresponders and will be included in the denominator when calculating ORR.

ORR and the corresponding 2-sided 90% exact CIs based on Clopper-Pearson method will be presented. A by-subject listing of overall response will be provided.

# 6.4.2. Time to Clinical Response CCI per Clinical Response Assessment

Time to clinical response in months will be calculated by (date of first clinical response - date of first dose of study drug + 1)/30.4375.

Time to clinical response will be summarized using descriptive statistics. A by-subject listing of time to clinical response will be provided.





For missing or incomplete dates of new anti-cancer therapy and death, imputation rules are described in Sections 6.3.2 and 6.3.1, respectively.



### 7. SAFETY ANALYSES

#### 7.1. Adverse Events and Deaths

# 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using the current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

### 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1, 2, 3, 4, or 5 according to CTCAE Version 4.03. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

# 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE CRF to the question of "Related to Study Treatment GS-4059", "Related to Study Treatment Idelalisib", or "Related to Study Treatment Obinutuzumab". Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if the AEs met the definitions of SAEs that were specified in the study protocol. SAEs captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Pharmacovigilance and Epidemiology Department before data finalization.

# 7.1.5. Treatment-Emergent Adverse Events

### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
- Any AEs leading to discontinuation of study drug

# 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

In case when the AE onset date is incomplete and needs to be imputed, the following algorithm will be followed:

- If the day is missing but the month and year are available, then the imputed day will be the first day of the month or the first dosing date if they have the same month and year, whichever is later.
- If the day and month are missing but year is available, then the imputed day and month will be 01Jan or the first dosing date if they have the same year, whichever is later.

### 7.1.6. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the Safety Analysis Set.

# 7.1.6.1. Summaries of AE Incidence by Severity

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, HLT, PT, and treatment group. For the AE categories described below, summaries will be provided by SOC, PT, maximum severity, and treatment group:

- TEAEs
- TEAEs with Grade 3 or higher
- TEAEs related to tirabrutinib
- TEAEs related to idelalisib
- TEAEs related to obinutuzumab

- TEAEs related to tirabrutinib with Grade 3 or higher
- TEAEs related to idelalisib with Grade 3 or higher
- TEAEs related to obinutuzumab with Grade 3 or higher
- TE SAEs
- TE SAEs related to tirabrutinib
- TE SAEs related to idelalisib
- TE SAEs related to obinutuzumab
- TEAEs leading to discontinuation of tirabrutinib
- TEAEs leading to discontinuation of idelalisib
- TEAEs leading to discontinuation of obinutuzumab
- TEAEs leading to dose modification of tirabrutinib
- TEAEs leading to dose modification of idelalisib
- TEAEs leading to dose modification of obinutuzumab
- TEAEs leading to temporary interruption of tirabrutinib
- TEAEs leading to temporary interruption of idelalisib
- TEAEs leading to temporary interruption of obinutuzumab
- TEAEs leading to discontinuation of study
- TEAEs leading to death (note that the severity will not be shown as all the TEAEs are Grade 5)

A brief, high-level summary of AEs described above will be provided by treatment group and by the number and percentage of subjects who experienced the above AEs. This summary table will also include TEAEs with Grade 3 or 4 and all deaths.

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and then by PT in descending order of total frequency within each SOC. For summaries by severity, the most severe severity will be used for those AEs that occurred more than once in a given subject during the study.

In addition to the above summary tables, TEAEs, TEAEs of Grade 3 or higher, TE treatment-related AEs, and TE SAEs will be summarized by PT only in descending order of total frequency.

In addition, data listings will be provided for the following:

- All AEs, indicating whether the event is treatment emergent
- All AEs with Grade 3 or higher
- All SAEs
- All Deaths
- AEs leading to death
- AEs leading to discontinuation of study drug
- AEs leading to discontinuation of study

# 7.1.6.1.1. Summary of Deaths

A summary (number and percentage of subjects) of deaths will be provided by treatment group. The summary will include the following categories:

- All deaths
- Deaths within 30 days of the last dosing of study drug
- Deaths beyond 30 days of the last dosing of study drug

The attribution of death will also be summarized.

#### 7.1.7. Adverse Events of Interest

The treatment-emergent AEs of interest (AEI) include:

| AEI | Grouped Terms |
|---|---|
| Hemorrhage/Bleeding | MST-CT Bleeding/Haemorrhage (Appendix 4) |
| Infections | SOC: Infections and infestations |
| Hypersensitivity | MST-CT Hypersensitivity (Appendix 5) |
| Cytopenia | MST: Anemia-related events, leukopenias, neutropenia, thrombocytopenias (Appendix 6) |
| Cardiac Arrhythmias | MST-CT Cardiac arrhythmia and bradycardia_narrow (Appendix 7) |
| Diarrhoea | PT: Diarrhoea |
| Rash | MST-CT Rash - specific to ONC (Appendix 8) |

The following summaries will be provided for AEIs by SOC, PT, and maximum severity:

- A) TEAE
- B) TEAEs leading to dose modifications or temporary interruption of study drug
- C) TEAEs leading to discontinuation of study drug

A data listing of AEIs will be provided by alphabetic ascending order of AEI name, then by subject ID.

# 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data in Appendix 9 will be provided for the Safety Analysis Set and will include data collected up to the last dose of study drug plus 30 days for subjects who have permanently discontinued study drug. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7. Hemolized test results will not be included in the analysis, but they will be listed in by-subject laboratory listings.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, and coagulation, separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on CTCAE severity grade will be flagged in the data listings, as appropriate.

No formal statistical testing is planned.

### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for each laboratory test specified in the study protocol as follows:

- Baseline values
- Postbaseline maximum value
- Postbaseline minimum value
- Change and percentage change from baseline to postbaseline maximum value
- Change and percentage change from baseline to postbaseline minimum value

A baseline laboratory value will be defined as the last measurement obtained on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; StD values will be displayed to the reported number of digits plus 1.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

# 7.2.2. Graded Laboratory Values

CTCAE Version 4.03 will be used to assign toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately. Local labs will be graded based on the central lab normal ranges with in-house macro.

# 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

# 7.2.2.2. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Graded TE laboratory abnormalities
- TE Grade 3 or 4 laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing postbaseline values up to 30 days after last dosing date.

A by-subject listing of treatment-emergent laboratory abnormalities will be provided by subject ID number and visit in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades and abnormal flags displayed.

# 7.2.3. Liver-related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements:

- Aspartate aminotransferase (AST): (a) > 3 times of the upper limit of reference range (ULN);
   (b) > 5 x ULN; (c) > 10 x ULN; (d) > 20 x ULN
- Alanine aminotransferase (ALT): (a) > 3 x ULN; (b) > 5 x ULN; (c) > 10 x ULN;
   (d) > 20 x ULN

- AST or ALT: (a)  $> 3 \times \text{ULN}$ ; (b)  $> 5 \times \text{ULN}$ ; (c)  $> 10 \times \text{ULN}$ ; (d)  $> 20 \times \text{ULN}$
- Total bilirubin: > 2 x ULN
- Alkaline phosphatase (ALP) > 1.5 x ULN
- AST or ALT > 3 x ULN and total bilirubin: (a) > 1.5 x ULN; (b) > 2 x ULN

The summary will include data from all postbaseline visits up to 30 days after the last dose of study drug. For individual laboratory tests, subjects will be counted once based on the most severe postbaseline values. For both the composite endpoint of AST or ALT and total bilirubin, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the Safety Analysis Set who have nonmissing postbaseline values of all relevant tests at the same postbaseline visit date. A listing of subjects who met at least 1 of the above criteria will be provided.

#### 7.2.4. Shifts Relative to the Baseline Value

Shift tables will be presented by showing change in severity grade from baseline to the worst postbaseline grade up to 30 days after last dosing date. The percentage will be based on subjects with values available at both baseline and postbaseline.

# 7.3. Body Weight and Vital Signs

Body weight and vital signs are collected at screening and may be collected at unscheduled visits. Thus, only a by-subject listing of vital signs will be provided by subject ID number and time visit in chronological order.

#### 7.4. Prior and Concomitant Medications

Medications collected at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary.

#### 7.4.1. Prior Medications

Prior medications are defined as any medications taken before a subject took the first study drug.

Prior medications will be summarized by Anatomical Therapeutic Chemical (ATC) drug class Level 2 and preferred name using the number and percentage of subjects for each treatment group and overall. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered alphabetically by ATC medical class and then by preferred term in order of descending overall frequency within each ATC medical class. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medication with a start date prior to the first dosing date of study drug will be included in the prior medication summary regardless of when the stop date is. If a partial start date is entered the medication will be considered prior unless the month and year (if day is missing) or year (if day and month are missing) of the start date are after the first

dosing date. Medications with a completely missing start date will be included in the prior medication summary, unless otherwise specified.

Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

#### 7.4.2. Concomitant Medications

Concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) drug class Level 2 and preferred name using the number and percentage of subjects for each treatment group. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered alphabetically by ATC medical class and then by preferred term in descending overall frequency within each ATC medical class. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medications with a start date prior to or on the first dosing date of study drug and continued to be taken after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified.

Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

# 7.5. Electrocardiogram Results

Electrocardiogram (ECG) analysis results are intended to identify meaningful changes in the QT interval. If potential abnormalities of interest are identified, further analyses may be conducted. Summaries of investigator assessment of ECG readings and ECG data will be provided for the Safety Analysis Set. No formal statistical testing is planned.

### 7.5.1. Investigator Electrocardiogram Assessment

A shift table of the investigators' assessment of ECG results at worst outcome during study compared with baseline values will be presented by treatment group using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant; or
missing. The number and percentage of subjects in each cross-classification group of the shift table will be presented. Subjects with a missing value at baseline or postbaseline will not be included in the denominator for percentage calculation. No formal statistical testing is planned.

A by-subject listing for ECG assessment results will be provided by subject ID number and visit in chronological order.

#### 7.5.2. Corrected QT Intervals

The QT interval (measured in millisecond [msec]) is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The QT interval represents electrical depolarization and repolarization of the ventricles. The QT interval is affected by heart rate, and a number of methods have been proposed to correct QT for heart rate.

Corrected QT (QTc) intervals will be derived using Fridericia's correction (QTcF) as follows:

$$QTcF = \frac{QT}{\sqrt[3]{RR}}$$

where QT is measured in msec; RR = 60/Heart Rate (beats per min [bpm]) and RR is measured in seconds

The maximum postdose QTcF interval values obtained during the study will be summarized within the following categories:

- $\bullet$  > 450 msec
- > 480 msec
- > 500 msec

The maximum postdose change in QTcF interval values obtained during the study will also be summarized within the following categories:

- > 30 msec
- > 60 msec

#### 7.5.3. PR and QRS Intervals

The PR interval (measured in msec) is a measure of the time between the start of the P wave (the onset of atrial depolarization) and the beginning of the QRS complex (the onset of ventricular depolarization). The QRS interval measures the duration of the QRS complex. The maximum ventricular rate (VR) and PR and QRS intervals observed during the study will be categorized. The number and percentage of subjects having values in the following ranges will be presented by treatment group:

• VR > 100 bpm

- PR interval > 200 msec
- QRS interval > 110 msec

### 7.6. Other Safety Measures

No additional safety measures are specified in the protocol.

### 7.7. Changes From Protocol-Specified Safety Analyses

There are no deviations from the protocol-specified safety analyses.



### 9. REFERENCES

Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, et al. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) updating the National Cancer Institute-Working Group (NCI-WG) 1996 guidelines. Blood 2008;111 (12):5446-56.

### 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

### 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| 16 Feb 2021 | 1 | Updated the protocol amendment number and date | To align with the latest protocol |
| 16 Feb 2021 | 4.4 | Added the section to provide how to handle special situations due to COVID-19 in the analysis | To assess the COVID-19 impact |
| 16 Feb 2021 | 5.3 | Revised the calculation of time since CLL diagnosis | To be consistent with the calculations of similar times |

### 12. APPENDICES

| Appendix 1. | Schedule of Assessments |
|-------------|--------------------------------------------------------|
| Appendix 2. | COVID-19 SMQ with Broad Scope |
| Appendix 3. | Determining Missing and Virtual Visits Due to COVID-19 |
| Appendix 4. | Bleeding/Haemorrhage Medical Search Term |
| Appendix 5. | Hypersensitivity Medical Search Term |
| Appendix 6. | Cytopenia Medical Search Term |
| Appendix 7. | Cardiac arrhythmia Medical Search Term |
| Appendix 8. | Rash Medical Search Term |
| Appendix 9. | List of Laboratory Tests for Safety Summary |

### **Appendix 1.** Schedule of Assessments

| | Screening | | | | | | | 24 V | Veeks | | | | | | | | | Every | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day -28 | 1 | Week<br>2<br>Day 1 | 3 | Week<br>4<br>Day<br>1 <sup>18</sup> | Week<br>5 | 7 | Week<br>9<br>Day 1 | 11 | 13 | 15 | Week<br>17<br>Day 1 | 19 | Week<br>21<br>Day 1 | Week<br>23 Day<br>1 | Week<br>25<br>Day 1 <sup>21</sup> | Week<br>29<br>Day 1 | 12 weeks<br>starting<br>Week 33<br>until<br>Week 105 | EOT <sup>19</sup> |
| Visit Window<br>(days) | | 0 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±7 | ±7 | ±7 | ±7 |
| Informed Consent | X | | | | | | | | | | | | | | | | | | |
| Medical and<br>Medication History <sup>1</sup> | X | | | | | | | | | | | | | | | | | | |
| Physical<br>Examination <sup>2</sup> | X | X | X | X | X | X | | X | | X | | X | | X | | X | X | X | X |
| Vital Signs | X | X | X | X | X | X | | X | | X | | X | | X | | X | X | X | X |
| ECOG Performance<br>Status / B-symptoms | X | X | | | | X | | X | | X | | X | | X | | X | X | X | X |
| Binet/Rai Staging | X | | | | | | | | | | | | | | | | | | |
| G8 Screening<br>Questionnaire <sup>3</sup> | | X | | | | | | | | | | | | | | X | | X | X |
| 12-lead ECG <sup>4</sup> | X | X | | | | X | | X | | X | | X | | X | | X | | | X |
| Adverse events/<br>Concomitant<br>medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tirabrutinib + idelalisib Dispensing <sup>5</sup> | | X | | | | X | | X | | X | | X | | X | | X | X | X | |
| Tirabrutinib + idelalisib Accountability | | | | | | X | | X | | X | | X | | X | | X | X | X | X |
| Obinutuzumab<br>Administration <sup>6</sup> | | X | X | X | | X | | X | | X | | X | | X | | | | | |
| Hematology <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Chemistry <sup>20</sup> | X | X | X | X | X | X | X | X | X | X | | X | | X | | X | X | X | X |


| | Screening | | | | | | | 24 V | Weeks | | | | | | | | | Every | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day -28 | 1 | Week<br>2<br>Day 1 | 3 | Week<br>4<br>Day<br>1 <sup>18</sup> | 5 | 7 | 9 | 11 | 13 | 15 | Week<br>17<br>Day 1 | Week<br>19<br>Day 1 | Week<br>21<br>Day 1 | Week<br>23 Day<br>1 | Week<br>25<br>Day 1 <sup>21</sup> | Week<br>29<br>Day 1 | 12 weeks<br>starting<br>Week 33<br>until<br>Week 105 | EOT <sup>19</sup> |
| Visit Window (days) | | 0 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±2 | ±7 | ±7 | ±7 | ±7 |
| Coagulation<br>(PT/INR, aPTT) | X | | | | | | | | | | | | | | | | | | X |
| Peripheral Blood<br>MRD <sup>8</sup> | | X | | | | | | | | X | | | | | | X | | X | X |
| Urinalysis and Urine<br>Chemistry | X | | | | | | | | | | | | | | | | | | |
| Pregnancy Testing <sup>9</sup> | X | X | | | | X | | X | | X | | X | | X | | X | X | X | X |
| Viral Serologies <sup>10</sup> | X | | | | | | | | | | | | | | | | | | |
| CMV Surveillance <sup>11</sup> | X | X | | | | X | | X | | X | | X | | X | | X | X | X | |
| CCI | | | | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | | | | |
| CLL phenotyping <sup>14</sup> | X | | | | | | | | | | | | | | | | | | X |
| Radiographic Tumor evaluation <sup>15</sup> | X | | | | | | | | | | | | | | | X | | | |
| Bone marrow evaluation <sup>16</sup> | X | | | | | | | | | | | | | | | X | | | |
| Response<br>Assessment <sup>17</sup> | | | | | | X | | X | | X | | X | | X | _ | X | X | X | X |

<sup>1</sup> Medical history includes significant past medical events (eg, prior hospitalizations or surgeries), a review of the disease under study, prior anti-cancer therapies, and any concurrent medical illnesses. CIRS score should be determined at screening.


<sup>2</sup> Screening and End of Treatment will be complete physical examinations. Beginning at Week 1 Day 1, a modified physical examination will be a performed to monitor for any changes (eg, lymph nodes, size of the liver and spleen, lung, cardiac, abdomen, skin, neurologic, and any system clinically indicated). Weight should be measured at screening only.

The G8 screening questionnaire will be used for assessment of subjects aged > 70 years at Week 1 Day 1 and every 6 months until EOT.

<sup>4</sup> Subjects should be resting quietly in supine position for 5 minutes prior to ECG collection. The Investigator or qualified designee will review all ECGs.

<sup>5</sup> Study drug is not dispensed at the Week 105 visit.

- 6 Obinutuzumab: 100 mg will be administered intravenously on Day 1 and 900 mg on either Day 1 or 2 (Week 1); then 1000 mg on Day 8 (Week 2), Day 15 (Week 3), and on Weeks 5, 9, 13, 17 and 21 for a total of 8 doses of 1000 mg over 21 weeks. If the 100 mg infusion on Day 1 is well tolerated, the remaining 900 mg (scheduled for Day 2) may be given on Day 1.
- 7 CBC with differential should be obtained every 2 weeks through Week 25 to evaluate for neutropenia and then at subsequent visits for assessment.
- 8 Peripheral blood MRD will be assessed on Day 1 of Weeks 1, 13, 25, 33, 45, 105, and EOT. EOT collection is not needed for subjects who complete the Week 105 visit.
- 9 Serum pregnancy test will be performed at screening for all women of childbearing potential. Urine pregnancy tests will be conducted prior to Week 1, Day 1 and then every 4 weeks until the EOT visit. Pregnancy kits may be provided for home testing The results must be confirmed as negative prior to continued administration of study drug.
- 10 Hepatitis serology includes HBsAg, HBcAb, HCV Ab; patients with positive HBcAb and negative HBsAg should have HBV DNA PCR performed prior to treatment start to rule out occult infection, then monthly through 6 months and then at subsequent clinic visits until EOT visit. HIV testing and CMV IgG and IgM testing should be performed at screening.
- 11 CMV antigen or quantitative PCR testing should be performed at screening and according to the schedule of assessments throughout the course of idelalisib treatment.
- CCI
- 14 CLL immunophenotyping, karyotyping and FISH, TP53 and IgHV mutation status, CD38 and ZAP70 expression will be evaluated from peripheral blood at screening. In the event of disease progression, only FISH and TP53 will be evaluated.
- 15 Tumor evaluation by CT scan (preferred) or MRI of neck, chest, abdomen, and pelvis will be performed at screening (unless scan was already completed up to 42 days prior to first dose). At the Week 25 visit, the same type of evaluation should be performed on those body regions which showed involvement by CLL at screening. An additional CT may be obtained on protocol per investigator discretion following evidence of an improvement in clinical response if the response assessment at the Week 25 visit is less than a complete response or in the event of suspected disease progression.
- A bone marrow evaluation is required in the screening window for subjects without radiographic evidence of disease. Bone marrow aspirate and biopsy should be performed at Week 25 for subjects fulfilling clinical response criteria for CR or CRi per the modified IWCLL 2008 criteria. MRD should be assessed from bone marrow aspirate at the reference laboratory in Kiel;
- CC
- Qualitative treatment response assessment based on physical exam, laboratory parameters and presence of B-symptoms should be performed every 4 weeks until Week 33 Day 1 and then at all scheduled visits thereafter following the modified IWCLL 2008 criteria, with the exception of lymphadenopathy, hepatomegaly, splenomegaly, and bone marrow. Assessment of response per modified IWCLL 2008 criteria should also be recorded at the completion of 24 weeks on treatment and subsequent to any CT and/or bone marrow biopsy that is repeated while on study.
- 18 Following evaluation of the safety data for the first 6 subjects enrolled in each treatment arm, the Safety Review Team (SRT) will determine if weekly clinical evaluation should continue for the duration of the study.
- 19 The EOT visit should be scheduled for approximately 30 days following discontinuation of all study treatment. For subjects that permanently discontinue all treatment prior to Week 25 Day 1, the Week 25 Day 1 visit should also be performed and may satisfy the requirement for the EOT visit if falling into the +30 days ± 7 day window from all study drug discontinuation.
- 20 Screening results should include creatinine clearance, serum thymidine kinase, serum beta2-microglobulin and serum quantitative immunoglobulins.
- 21 The window for bone marrow assessments is -7 days or +14 days as calculated from Week 1 Day 1.


### Appendix 2. COVID-19 SMQ with Broad Scope

Note: The list presented below is based on MedDRA Version 23.1. The actual list will be up-versioned to the MedDRA version used at the time of database finalization.


#### Appendix 3. Determining Missing and Virtual Visits Due to COVID-19

This appendix describes the clinical trial site collection of COVID-19 data pertaining to missed/virtual visits and the data processing algorithm used to determine which visits were missing and which visits were virtual.

#### Data collection

A COVID-19 supplement to the eCRF Completion Guidelines (CCG) was provided by data management to instruct clinical trial sites with respect to data entry expectations pertaining to scenarios related to the COVID-19 pandemic. If a visit was missed, sites should enter "Visit missed due to COVID-19." If an in-person visit was conducted virtually, sites should enter "Virtual visit due to COVID-19."

#### Determination of Missed and Virtual visits

NLP was used to search the CRF comment fields to identify instances of "COVID-19" (or synonyms, see the table below) and "Virtual" (or synonyms, see the table below). The search terms are maintained in a global lookup table and can be modified to tune the NLP model. For any comments with COVID-19 search terms, assign "Missed visit" or "Virtual visit as follows:

- i. If COVID-19 terms are identified through NLP and the visit date is missing, then result is "Missed Visit"
- ii. If COVID-19 and Virtual terms are identified through NLP for a visit, then result is "Virtual Visit". When there are multiple records for the same subject and the same visit, NLP will be based on multiple records to ensure 1 unique category per subject per visit
- iii. Otherwise result is missing

# Examples of Search Terms for "COVID-19" and "Virtual" Used to Identify Missed and Virtual Visits

| Search Terms for "COVID-19" | Search Terms for "Virtual" |
|-----------------------------|----------------------------|
| COVID19 | VIRTUAL |
| CORONA | TELEMED |
| CORONAVIRUS | TELEHEALTH |
| PANDEMIC | TELEPHONE |
| OUTBREAK | REMOTE |
| CRISIS | TELEMEDICINE |
| LOCKDOWN | TELECONSULTATION |
| QUARANTINE | TELEPHONICALLY |
| SHELTER | PHONE |
| | HOME VISIT |
| | ZOOM |
| | SKYPE |

### Appendix 4. Bleeding/Haemorrhage Medical Search Term

Note: The list presented below is based on MedDRA Version 22.0. The actual list will be up-versioned to the MedDRA version used at the time of database finalization.


### Appendix 5. Hypersensitivity Medical Search Term

Note: The list presented below is based on a SMQ in MedDRA Version 22.0. The actual list will be up-versioned to the MedDRA version used at the time of database finalization.


### Appendix 6. Cytopenia Medical Search Term

Note: The list presented below is based on MedDRA Version 22.0. The actual list will be upversioned to the MedDRA version used at the time of database finalization.


### Appendix 7. Cardiac arrhythmia Medical Search Term

Note: The list presented below is based on MedDRA Version 22.0. The actual list will be upversioned to the MedDRA version used at the time of database finalization.


### **Appendix 8.** Rash Medical Search Term

Note: The list presented below is based on MedDRA Version 22.0. The actual list will be upversioned to the MedDRA version used at the time of database finalization.


### **Appendix 9.** List of Laboratory Tests for Safety Summary

| Serum Chemistry | Hematology |
|---|---|
| Sodium Potassium Chloride Glucose Blood urea nitrogen or urea Creatininea ALT AST GGT Cholesterol Triglycerides Uric Acid | WBC RBC Hemoglobin Hematocrit Platelet Count Neutrophils (ANC) Lymphocytes Monocytes Basophils Eosinophils |
| Alkaline phosphatase Total and direct bilirubin | Coagulation |
| Total protein Albumin Calcium Magnesium Phosphate LDH | PT/INR<br>aPTT |

a Estimated creatinine clearance/glomerular filtration rate will be calculated based on the Cockroft-Gault formula ALT = alanine aminotransferase; aPTT = activated partial thromboplastin time; AST = aspartate aminotransferase; BUN = blood urea nitrogen; GGT = gamma-glutamyltransferase; INR = international normalized ratio; LDH = lactate dehydrogenase; PT = prothrombin time; RBC = red blood cell; WBC = white blood cell

## GS-US-401-1958 SAP V2.0

### **ELECTRONIC SIGNATURES**

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:mm:ss) |
|---|---|---|
| PPD | Clinical Research eSigned | 16-Feb-2021<br>23:09:33 |
| PPD | Biostatistics eSigned | 19-Feb-2021<br>06:56:57 |